CLINICAL TRIAL: NCT00812383
Title: Carotid With Bivalirudin Angioplasty
Acronym: COBRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COBRA
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Carotid Artery Disease
MeSH Terms: conditions — Carotid Artery Diseases

ARMS (2):
- Bivalirudin (Experimental)
  Interventions: Device: RX ACCULINK™ Carotid Stent System; RX ACCUNET™ Embolic Protection System; PercuSurge GuardWire® 3-6 Temporary Occlusion and Aspiration System
- Heparin (Active Comparator)
  Interventions: Device: RX ACCULINK™ Carotid Stent System; RX ACCUNET™ Embolic Protection System; PercuSurge GuardWire® 3-6 Temporary Occlusion and Aspiration System

INTERVENTIONS:
Device: RX ACCULINK™ Carotid Stent System; RX ACCUNET™ Embolic Protection System; PercuSurge GuardWire® 3-6 Temporary Occlusion and Aspiration System — Angiomax (bivalirudin) versus standard anticoagulation with heparin during carotid artery stenting with distal protection clinical endpoint evaluation

SUMMARY:
Single center randomized clinical trial, to evaluate the safety and efficacy of carotid artery stenting using the RX ACCULINK™ Carotid Stent System with RX ACCUNET™ Embolic Protection System or PercuSurge GuardWire® 3-6 Temporary Occlusion and Aspiration System using Angiomax (bivalirudin)versus heparin as the anticoagulant for treatment of occlusive carotid artery disease in low and high risk patient cohorts.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age.
* The patient must have a significant diameter reduction of the extracranial or intracranial internal or common carotid artery, defined as ≥50% stenosis for symptomatic patients or ≥80% stenosis for asymptomatic patients determined by carotid duplex ultrasound scan and/or carotid angiography.
* Female patients with child bearing potential must have a negative pregnancy test.
* The patient and the patient's physician must agree to have the patient return for a 30-day and one-year clinical and ultrasound imaging follow-up evaluations as indicated in the protocol.
* Reference vessel diameter ≥ 3.5 mm - ≤ 9.0 mm diameter.

Exclusion Criteria:

* The patient has had a recent (<4 weeks) disabling stroke or dementia with major neurologic deficit (stroke scales: Barthel <60, NIH >15, or Rankin >3) at pre-procedure neuro exam.
* The patient has had within four weeks of the treatment procedure an intracranial hemorrhage, hemorrhage stroke, major stroke, or any stroke with mass effect demonstrated on MRI or CT.
* The patient has a known allergy to heparin, bivalirudin, aspirin or to anti-platelet agents that prevents taking aspirin plus ticlopidine or aspirin plus clopidogrel.
* The patient has received fractionated or unfractionated heparin within 8 hours prior to the procedure.
* The patient has a history of prior life-threatening radiocontrast reaction that cannot be pre-treated.
* The patient has a history of bleeding diathesis or coagulopathy within 3 months.
* The patient is currently participating in another study protocol that may influence either procedure results or follow-up evaluations.
* Plasma/serum creatinine > 3.0 mg/dl at time of intervention.
* Hemodynamic instability at the time of intervention.
* Previous stent placement in the ipsilateral carotid distribution.

Angiographic Exclusion Criteria

* The patient has an intracranial tumor, or cerebral arterio-venous malformation(s) > 5mm, aneurysms or severe intracranial stenosis distal to target lesion.
* The patient has inaccessible intracranial arterial stenosis greater in severity than the extracranial internal carotid artery lesion.
* There is angiographic evidence of significant intra-luminal thrombus burden with presumed increased risk of plaque fragmentation and consequent distal embolization.
* There is total occlusion of the ipsilateral carotid artery treatment site with TIMI 0 flow characteristics.
* The reference segment diameter (internal carotid artery segment cephalad to the lesion) is less than 3 millimeters by operator visual estimate.
* The patient has peripheral vascular, supra-aortic or internal carotid artery tortuosity precluding use of catheter-based techniques required for successful CSSA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
To evaluate clinical success (<50% residual stenosis at all treatment sites without death, myocardial infarction, stroke or major bleed) | 30 days

SECONDARY OUTCOMES:
To assess for complications including death, myocardial infarction, major or minor stroke, major or minor bleeding, and vascular complications. | In hospital and 30 days
To assess stent patency , and occurence of death or recurrent neurological events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lowell Satler, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States